CLINICAL TRIAL: NCT01820663
Title: Dietary Intervention in Stroke Recovery in the Acute Rehabilitation Setting With the Modified Atkins Diet.
Brief Title: Dietary Intervention With the Modified Atkins Diet in Stroke Rehabilitation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Burke Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Carolin Dohle, Neurology Attending, Burke Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BRH-424
Record Dates: First submitted 2013-03-13; First posted 2013-03-29 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Stroke; Ischemic Stroke
Keywords: stroke; ketones; ketogenic diet; impairment; disability
MeSH Terms: conditions — Stroke; Ischemic Stroke; Ketosis | interventions — Diet, Sodium-Restricted; Diet; Diet, Diabetic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Modified Atkins Diet (Experimental): Patients will receive a 14 day menu consisting of the Modified Atkins diet, a low-carbohydrate, high protein, high fat diet.
  Interventions: Other: Modified Atkins Diet
- Control Diet (Placebo Comparator): Patients will receive a diet (e.g. regular, low cholesterol, diabetic) determined by the attending physician.
  Interventions: Other: Control diet

INTERVENTIONS:
Other: Modified Atkins Diet — A high fat, high protein, low- carbohydrate diet
  Arms: Modified Atkins Diet
Other: Control diet — The control diet is a diet determined by the attending physician caring for the patient and may consist of either a low sodium diet, a low sodium/ low cholesterol diet, a regular diet or a diabetic diet.
  Other Names: Low sodium diet; low sodium/ low cholesterol diet; regular diet; diabetic diet
  Arms: Control Diet

SUMMARY:
This phase 1 study tests whether use of the Modified Atkins Diet (MAD) can improve motor impairment after stroke. It is based on the hypothesis that after stroke, the brain's utilization of glucose, it's primary source of energy, is disrupted. The MAD is a low-carbohydrate diet that has can switch the body's metabolism from using glucose to using products of fat metabolism, so-called ketones. Ketones may act as an alternative energy substrate for the brain. Ketones also have several neuroprotective effects after stroke.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-99
* First time unilateral hemispheric ischemic stroke. Not more than 12 weeks after acute stroke.
* Burke Stroke Rehabilitation Unit Inpatient.
* Preserved cognitive ability to understand commands and participate in outcome measures and to give informed consent. In patients with aphasia, cognitive ability to give consent will be determined by a physician.
* Upper extremity motor impairment with an UE Fugl Meyer score ≤ 56/66
* Independence in ADLS/ absence of major impairment prior to stroke

Exclusion Criteria:

* Hemorrhagic stroke
* Uncontrolled hyperlipidemia with LDL > 250 on admission
* Uncontrolled Diabetes mellitus with BS > 300 averaged over the first day of admission
* Nutritional risk as defined by BMI < 18.5 or by a score of 2 or higher on the Malnutrition Universal Screening Tool (scores BMI, % of unplanned weight loss in last 3-6 months and question whether patient is acutely ill)
* Decreased renal function with eGFR <30%
* Stage III and IV pressure ulcers
* Osteoporosis not sufficiently treated with oral Calcium and Vitamin D supplements
* CHF as defined by class III or worse
* Hypersensitivity/allergy to cholesterol lowering medications
* H/o kidney stones within last 1 year prior to stroke or medications predisposing to kidney stones such as Topamax, carboanhydrase inhibitors
* Inability to tolerate an oral diet and need for tube feeds
* Active enrollment in any other interventional studies at Burke; enrollment in observational studies or studies using TMS as a measurement may not pose exclusion criteria
* Cognitively unable to follow instructions.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change in Upper Extremity Fugl Meyer Motor Score | assessed upon beginning of the study, discharge from Burke Rehabilitation Hospital (average 25 days post study enrollment) and at 3 months post discharge
  The Upper Extremity Fugl Meyer Motor Score is used to assess impairment in upper extremity function. Individuals are asked to complete a certain sequence of movements, and quality of movements is scored.

SECONDARY OUTCOMES:
Change in Montreal Cognitive Assessment (MOCA) | assessed upon beginning of the study, discharge from Burke Rehabilitation Hospital (average 25 days post study enrollment) and at 3 months post discharge
  The MOCA is an assessment of cognitive impairment and evaluates several cognitive domains.

CONTACTS AND LOCATIONS:
Overall Officials: Carolin I Dohle, MD, Principal Investigator — Burke Rehabilitation Hospital
Locations (1):
- Burke Rehabilitation Hospital, White Plains, New York, United States

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be disclosed.